CLINICAL TRIAL: NCT05320081
Title: Camrelizumab Combined With CD30 CAR-T in the Treatment of Relapsed/Refractory CD30+ Lymphoma: a Single-arm, Open-label Clinical Study
Brief Title: Camrelizumab Combined With CD30 CAR-T in the Treatment of Relapsed/Refractory CD30+ Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Jianfeng Zhou, Director of the Division of Hematology, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-ML-Ⅱ-001
Record Dates: First submitted 2021-11-24; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Lymphoma; Relapse/Recurrence
Keywords: CD30 positive
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with CD30 CAR-T (Experimental): This study have only one arm that is Camrelizumab combined with CD30 CAR-T experimental arm.
  Interventions: Biological: CD30 CAR-T; Drug: Camrelizumab

INTERVENTIONS:
Biological: CD30 CAR-T — Subjects need to complete a series of checks before reinfusion of CD30 CAR-T cells as baseline information for subjects after non-myeloablative pretreatment. The subject was reinfused with CD30 CAR-T cells (10±3)×10^6/kg on the 0th day of the first dosing cycle (the investigator decided the specific reinfusion dose based on the subject's own/disease conditions and preparation conditions in vitro ), concurrent oxygen inhalation and monitoring (ECG, blood pressure and blood oxygen monitoring). The reinfusion was completed in about 30 minutes, and the tube was flushed with saline.
  Note: CAR-T cell infusion and reinfusion dose are based on the subject's condition.
Drug: Camrelizumab — Received Camrelizumab treatment on the 15th day after CAR-T cell reinfusion, and then received Camrelizumab treatment every 2 weeks.

SUMMARY:
The is a phase II, single-arm, open-label clinical study assessing the efficacy and safety of Camrelizumab combined with CD30 CAR-T in the treatment of r/r CD30+ lymphoma. Plan to recruit 30 subjects with r/r CD30+ lymphoma。

DETAILED DESCRIPTION:
This study intends to combine CD30 CAR-T (provided by Wuhan Bio-Raid Biotechnology Co., Ltd) and Camrelizumab (provided by Jiangsu Hengrui Pharmaceutical Co., Ltd.) to treat r/r CD30+ lymphoma, to observe the safety and effectiveness of the combined treatment, and to study the effect of PD-1 antibody on the pharmacokinetics and pharmacodynamics of CAR-T. Obtain a better treatment plan and provide a new strategy for the treatment of clinically r/r CD30+ lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years and ≤70 years，female and male；
* ECOG performance status 0-2；
* Histological or flow cytometry confirmed CD30+ lymphoma [according to WHO2008 diagnostic standard]
* Patients with CD30+ lymphoma relapsed after ≥2 lines of systemic treatment (the disease progresses after treatment remission) or refractory ( failed to obtain CR after previous systemic treatment)；
* The patient did not receive any chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs) and other anti-cancer treatments within 4 weeks before enrollment, and the treatment-related toxicity has recovered to ≤ Grade 1 (except for alopecia) 4 weeks before enrollment；
* At least 1 evaluable or measurable lesion can be measured according to the LYRIC 2016 evaluation criteria for malignant lymphoma ；
* Sufficient organ and bone marrow function, no serious abnormalities neither in hematopoietic function nor in heart, lung, liver, and kidney functions, and no immune deficiencies;

  1. The absolute value of neutrophils is ≥1.5×109/L (for patients with bone marrow invasion ≥1.0×109/L);
  2. Platelets ≥75×109/L (patients with bone marrow invasion ≥50×109/L);
  3. Hemoglobin ≥9 g/dL;
  4. Serum creatinine ≤ 1.5× the upper limit of normal (ULN), or creatinine clearance ≥40 mL/min (estimated based on the Cockcroft-Gault formula);
  5. Serum total bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN ( liver invasion);.
  6. f) Aspartate aminotransferase、Alanine Aminotransferase (ALT) ≤2.5 × ULN or ≤5 × ULN ( liver invasion);
  7. Coagulation function: International Normalized Ratio (INR) ≤ 1.5 × ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN (the PT and APTT should be within the expected range of anticoagulant therapy at the time of screening if the subject is receiving anticoagulant therapy,).
  8. Thyroid-stimulating hormone (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) are within ±10% of the normal value.
  9. Left ventricular ejection fraction (LVEF) ≥ 50%, no serious malignant arrhythmia;
* The estimated survival time ≥6 months;
* Sufficient understanding and voluntarily to sign the informed consent form;
* Patients with fertility must be willing to be able to use reliable contraceptive measures during the clinical study and within 12 months after the last administration

Exclusion Criteria:

* Lymphoma associated hemophagocytic syndrome;
* Patients diagnosed as primary cutaneous anaplastic large cell lymphoma （ALCL） (patients can be enrolled if ALCL is transformed from other organ involvement);
* Patients with malignant T cells involving bone marrow or peripheral blood;
* Suffered from other malignant tumors in the past 5 years, except for for skin basal cell carcinoma, skin squamous cell carcinoma, breast carcinoma in situ and cervical carcinoma in situ undergoing the radical treatment
* Received CAR-T therapy or other genetically modified cell therapy before screening
* Received other treatments that affect the collection of T cells for when enrolled or within 4 weeks before enrollment;
* Suffer from active autoimmune diseases that require systemic treatment in the past two years (hormone replacement therapy is not considered as systemic treatment, such as type I diabetes, hypothyroidism that requires only thyroxine replacement therapy, patients with low adrenal function or hypopituitarism who need only physiological doses of glucocorticoid replacement therapy);
* Patients with uncontrolled infectious diseases, active viral hepatitis, tuberculosis, and HIV-infected ;
* Known to be allergic to ampicillin, antibodies, cytokines, anti-PD-1/PD-L1 antibodies or pharmaceutical excipients; or have severe allergic reactions to other monoclonal antibodies;
* Previous use of immunosuppressive drugs within 14 days before the first use of the drug, excluding nasal sprays and inhaled corticosteroids or physiological doses of systemic steroid hormones (ie not more than 10 mg/day prednisolone or equivalent physiological doses of other corticosteroids);
* long-term use of systemic hormones (dose equivalent to >10mg prednisone/day) or any other form of immunosuppressive therapy is required. Subjects using inhaled or topical corticosteroids can be enrolled;
* Suffer from uncontrolled comorbidities, including but not limited to symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer or bleeding disorders.
* With history of interstitial lung disease or non-infectious pneumonia. Subjects who have previously had drug-induced or radioactive non-infectious pneumonia but asymptomatic are allowed to enroll.
* Patients have other conditions that are not suitable for enrollment according to the judgment of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | up to 3 months after CAR-T cell infusion
  including complete remission (CR) or partial remission (PR)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 90 days
  To evaluate the safety of camrelizumab combined with CD30 CAR-T in the treatment of relapsed/refractory CD30+ lymphoma.

SECONDARY OUTCOMES:
overall survival (OS) | 24 months
  The time from the day of enrollment to death due to any cause. If it is unclear whether the subject has died, OS refers to the duration from the day of enrollment to the date of the last follow-up.
Duration of remission (DOR) | 24 months
  Defined as the time between the initial appearance of complete or partial remission for a subject in objective remission to the appearance of disease recurrence or death from any cause (whichever occurs first).
Progression-free Survival (PFS) | 24 months
  The time from the start of the trial to the day of PD or to death due to any reason. If the subject's disease status is unclear, PFS refers to the duration from the day of enrollment to the date of the last follow-up.
Time to Remission (TTR). | 12 months
  The time from the first day of medication to the first assessment of PR or CR, whichever comes first. Only applicable to subjects with CR or PR.

OTHER OUTCOMES:
The copy number of CD30 CAR-T cells | 12 months
  The copy number of CD30 CAR-T cells amplified (copies/mcgDNA) in peripheral blood after administration;

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhou, Principal Investigator — Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Department of Hematology Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No